CLINICAL TRIAL: NCT01342783
Title: Next Generation Sequencing of Childhood Soft Tissue Sarcomas to Identify Drivers of Primary and Metastatic Disease
Brief Title: Biomarkers in Samples From Young Patients With Soft Tissue Sarcoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ARST11B2; COG-ARST11B2 (Other: Children's Oncology Group); NCI-2011-02853 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ARST11B2 (Other: Children's Oncology Group)
Record Dates: First submitted 2011-04-23; First posted 2011-04-27 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Sarcoma
Keywords: metastatic childhood soft tissue sarcoma; nonmetastatic childhood soft tissue sarcoma; recurrent childhood soft tissue sarcoma; previously treated childhood rhabdomyosarcoma; previously untreated childhood rhabdomyosarcoma; recurrent childhood rhabdomyosarcoma
MeSH Terms: conditions — Sarcoma | interventions — Base Sequence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA analysis
Genetic: RNA analysis
Genetic: mutation analysis
Genetic: nucleic acid sequencing
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer.

PURPOSE: This research trial is studying biomarkers in samples from young patients with soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify the key components of driver pathways of primary and secondary soft tissue sarcomas.
* To perform the next-generation sequencing on primary versus normal on undifferentiated sarcomas.

OUTLINE: Genomic DNA and RNA samples from undifferentiated sarcoma tumors are analyzed by next-generation sequencing for somatic mutations. Normal matched lymphocytes and tissue are also analyzed.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Banked childhood samples from the COG-D9902 soft tissue sarcoma biology and banking study
* Rhabdomyosarcoma, NOS

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: COG-D9902 soft tissue sarcoma biology and banking study participants.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-05; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of somatic mutations in driver genes and mutations in other genes that occur individually

CONTACTS AND LOCATIONS:
Overall Officials: Poul Sorensen, MD, PhD, Principal Investigator — British Columbia Cancer Agency